CLINICAL TRIAL: NCT01156857
Title: A Phase III, Multicentre, Clinical Study Investigating the Efficacy and Safety of 3-months Open-label Treatment With PGL4001, Followed by a Randomised, Double-blind Placebo Controlled Period of 10 Days Treatment With Progestin, in Subjects With Myomas and Heavy Uterine Bleeding.
Brief Title: PGL4001 Efficacy Assessment in Reduction of Symptoms Due to Uterine Leiomyomata
Acronym: PEARLIII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PregLem SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PGL09-026
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2013-06

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — ulipristal acetate; Progestins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Drug: PGL4001 10mg (oral tablets) for 3 months followed by a period of 10 days of placebo (oral tablets).
  Interventions: Drug: PGL4001, placebo
- B (Experimental): Drug: PGL4001 10mg (oral tablets) for 3 months followed by a period of 10 days of progestin (oral tablets).
  Interventions: Drug: PGL4001, progestin

INTERVENTIONS:
Drug: PGL4001, placebo — PGL4001 10mg once daily (oral tablets) for 3 months followed by a period of 10 days of placebo (oral tablets).
  Other Names: Ulipristal acetate
  Arms: A
Drug: PGL4001, progestin — PGL4001 10mg once daily (oral tablets) for 3 months followed by a period of 10 days of progestin Norethisterone acetate 10mg once daily (oral tablets).
  Other Names: Ulipristal acetate
  Arms: B

SUMMARY:
This is a multicentre, Phase III, efficacy and safety open-label study with PGL4001 10mg once daily for 3 months, blinded towards the administration of progestin or placebo after end of PGL4001 treatment.

DETAILED DESCRIPTION:
PGL4001 will be administered daily to all subjects in an open-label manner with no control group. The three months open label treatment period will be followed by a ten day double blind treatment with progestin or matching placebo. Subjects will be randomly assigned to progestin or matching placebo arm with a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a pre-menopausal woman aged between 18 and 48 years inclusive.
* Subject with a Body Mass Index ≥18 and ≤40.
* Subject with myomatous uterus size < 16 weeks.
* Subject must have at least one uterine myoma of at least 3 cm diameter in size and no myoma larger than 10 cm diameter diagnosed by ultrasound.
* Subject complained of strong uterine bleeding.
* Subject is eligible for hysterectomy or myomectomy.
* Females of childbearing potential have to practice a non-hormonal method of contraception.

Exclusion Criteria:

* Subject has a history of or current uterus, cervix, ovarian or breast cancer.
* Subject has a history of endometrium hyperplasia or adenocarcinoma in a biopsy performed within the past 6 months or similar lesions in the screening biopsy.
* Subject has a known severe coagulation disorder.
* Subject has a history of treatment for myoma with a SPRM, including ulipristal acetate.
* Subject has abnormal hepatic function at study entry.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2010-07; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Efficacy endpoints | From baseline to end of PGL4001 treatment (3months treatment) and to approximately 2 weeks after double blind treatment with progestin/placebo.
  Investigate efficacy of PGL4001 on uterine bleeding (% of subjects in amenorrhea at end of PGL4001 treatment), myoma size (transvaginal ultrasound), pain (short Mc Gill questionnaire) and quality of life (specific UFS-QoL questionnaire and general EQ-5D questionnaire).
Number and proportion of subjects experiencing open label treatment-emergent adverse events | From baseline to end of PGL4001 treatment (3months treatment)

CONTACTS AND LOCATIONS:
Locations (22):
- Austria (2):
  - Medical University Graz, department of obstetrics and gynecology, Graz
  - Medical University Vienna, department of obstetrics and gynecology, Vienna
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHR de la citadelle, Liège
  - Cliniques Universitaires UCL de Mont-Godinne, Yvoir
- Poland (8):
  - Prywatna Klinika Polozniczo-Ginekologiczna, Bialystok
  - INVICTA Sp. Z o.o., Gdansk
  - Private Practice, Katowice
  - Private Practice, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 w Lublinie Klinika Ginekologii Onkologicznej i Ginekologii, Lublin
  - Private Practice, Warsaw
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Klinika Poloznictwa, Chorob Kobiecych i Ginekologii Onkologicznej, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wrocławiu, I Katedra i Klinika Ginekologii i Położnictwa, Wroclaw
- Spain (9):
  - Institut Universitari Dexeus Departamento de Ginecología, Barcelona
  - Hospital Universitario Hebron, gynecology department, Barcelona
  - Hospital Clinic i provincial de Barcelona, gynecology department, Barcelona
  - Hospital General de Ciudad Real Gynecology, Ciudad Real
  - Hospital Universitario de Guadalajara Consultas de Ginecología (Planta 0), Guadalajara
  - Clinica Ginecologica CEOGA, departamento de Ginecologia, Lugo
  - Private pratice, Madrid
  - Hospital universitario 12 de Octubre, departamento de ginecologia, Madrid
  - CHIP, Málaga

REFERENCES:
- [Derived] Donnez J, Vazquez F, Tomaszewski J, Nouri K, Bouchard P, Fauser BC, Barlow DH, Palacios S, Donnez O, Bestel E, Osterloh I, Loumaye E; PEARL III and PEARL III Extension Study Group. Long-term treatment of uterine fibroids with ulipristal acetate ☆. Fertil Steril. 2014 Jun;101(6):1565-73.e1-18. doi: 10.1016/j.fertnstert.2014.02.008. Epub 2014 Mar 12. PMID 24630081